CLINICAL TRIAL: NCT05213520
Title: Effect of a Novel Alternate Day Intermittent Energy Restriction Intervention vs. Standard Reduced Calorie Diet on Body Weight, Body Composition, and Resting Metabolic Rate in College Students With Obesity
Brief Title: Effect of a 4-week Alternate Day Intermittent Energy Restriction Intervention vs Reduced
Acronym: AltER2022
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University (Other)
Responsible Party: Principal Investigator, Martin Binks, Professor, Texas Tech University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB2021-1092
Record Dates: First submitted 2022-01-18; First posted 2022-01-28 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2022-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: 30 participants will be randomized into 1 of 2 groups 1) n=15 the experimental group that will receive the alternate day intermittent energy restriction intervention and 2 n=15 will be active control group that will follow a standard reduced calorie diet.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alternate Day Intermittent Energy Restriction (Experimental): Participants assigned to this diet will be asked to alternate between full calorie (no restriction) eating days with eating 40% of their daily caloric requirement on the other day. For example, if their requirement is 2000 calories they would eat 800 calories one day and as much as you want on the other day and repeat every two days. There will be occasional exceptions allowed with maximum of two 40% days in a row (followed by two full days) based on personal schedule with prior approval. They will follow this for 4 weeks.
  Interventions: Other: Alternate Day Intermittent Energy Restriction
- Reduced Calorie Diet (Active Comparator): Participants assigned to this diet will be asked to restrict calorie intake by 500-1000 calories below their daily energy requirement every day. They will follow this for 4 weeks.
  Interventions: Other: Reduced Calorie Diet

INTERVENTIONS:
Other: Alternate Day Intermittent Energy Restriction — It is a dietary intervention designed to alternate between full energy consumption on one day and 40% of daily energy requirement on the following day.
  Arms: Alternate Day Intermittent Energy Restriction
Other: Reduced Calorie Diet — It is a dietary intervention designed to reduce daily calorie intake by 500-1000 kcal below an individual's daily calorie needs.
  Arms: Reduced Calorie Diet

SUMMARY:
This pilot study is an active control randomized controlled trial with a sample size of 30 that will consist of 2 groups, to evaluate the effects of a one-month alternate day intermittent energy restriction (AltER) intervention on body weight, body composition, resting metabolic rate in college students with obesity as compared to a standard reduced calorie diet (RCD). Among the 30 participants, 15 will be randomized into the experimental group that will receive the AltER intervention while the other 15 will be a part of the active control group that will follow a RCD. The study will be conducted at the Texas Tech University Nutrition and Metabolic Health Initiative.

DETAILED DESCRIPTION:
This pilot study proposes to investigate the scope and benefits of a novel, hybrid alternate day fasting protocol tailored to the college student lifestyle. This protocol - Alternate Day Intermittent Energy Restriction (AltER) is novel because it proposes to modify the standard ADF regime by increasing energy intake to 40% of calorie needs on fasting days. While this may not be as restrictive as other protocols, it still can help create a significant energy deficit. Additionally, it will provide flexibility by allowing for two consecutive fast days if the individual chooses to. While most dietary interventions can achieve significant weight loss in this short duration we expect that this approach tailored to college lifestyle will be superior to typical dietary restriction.

Subjects will be asked to attend two approximately 90-minute assessment visits (4 weeks apart) at the NMHI facility They will have their height weight and blood pressure measured, fill out questionnaires (attached), and have body composition (BodPod) and resting metabolic rate (Metabolic Cart) measured.

At completion of visit one they are randomly assigned to one of two Diet protocols designed to reduce calories and help them to safely lose weight They will also be asked to respond to a brief (3 questions) email survey weekly.

The AltER diet alternate between full calorie (no restriction) eating days with eating 40% of your daily caloric requirement on the other day. There will be occasional exceptions allowed with maximum of two 40% days in a row (followed by two full days) based on personal schedule with prior PI approval. The RCD will require a reduction of 500-1000 calories below daily energy requirement. The intervention or control diet will be followed for a duration of 4 weeks at the end of which the participants will come in for visit 2 which will follow a similar format like visit 1.

General Aim

To determine the effect of a novel, alternate day intermittent calorie restriction intervention on body weight, fat mass and resting metabolic rate of college students with obesity as compared to a standard reduced calorie diet 3.2.1. Specific Aim 1: To determine the effect of a novel, alternate day intermittent calorie restriction intervention on body weight of college students with obesity as compared to a standard reduced calorie diet.

3.2.1. Specific Aim 2: To determine the effect of a novel, alternate day intermittent calorie restriction intervention on fat mass of college students with obesity as compared to a standard reduced calorie diet.

3.2.2. Specific Aim 3: To determine the effect of a novel, alternate day intermittent calorie restriction intervention on resting metabolic rate of college students with obesity as compared to a standard reduced calorie diet.

3.2.2. Specific Aim 4: To explore the relationships of stress, sleep physical activity and weight history/demographic variables in relation to primary outcomes of interest.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 -25 years
2. Enrolled as full-time college students
3. Have a BMI ≥ 30
4. Willing and able to give informed consent
5. Willing to follow either dietary intervention assigned to them upon randomization.
6. Able to come in for all assessment visits.

Exclusion Criteria:

1. Participants who are currently diagnosed with diabetes mellitus, cardiovascular disease, liver or kidney disease, cancer
2. Current severe psychiatric illnesses (e.g. psychosis, schizophrenia, bipolar disorders, depression
3. Current suicidal ideation, and recent or past suicide attempts
4. History of psychiatric hospitalization (past year).
5. History of diagnosed eating disorders such as bulimia nervosa, anorexia nervosa and severe binge eating disorder.
6. History of diagnosed substance abuse or alcohol abuse.
7. Currently on any weight loss diet.
8. Having lost in the past 3 months 10% or more of body weight.
9. Unwilling or unable to give informed consent.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2022-01-13 (Actual); Primary Completion 2022-11-05 (Actual); Study Completion 2022-11-05 (Actual)

PRIMARY OUTCOMES:
Body Weight | 4 weeks
  Change in body weight in pounds.
Fat Mass | 4 weeks
  Change in fat mass in pounds as measured by body composition assessment.
Resting Metabolic Rate | 4 week
  Change in resting metabolic rate as measured by indirect calorimetry.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Binks, Ph.D., Principal Investigator — Texas Tech University- Department of Nutritional Sciences
Locations (2):
- United States (2):
  - Texas Tech University - Department of Nutritional Sciences, Lubbock, Texas
  - Nutrition and Metabolic Health Initiative, Lubbock, Texas

IPD SHARING:
Plan to Share IPD: No